CLINICAL TRIAL: NCT04999488
Title: Impact of Orally Administered BPM31510 on Mitochondrial Energetics in Older
Brief Title: Impact of Orally Administered BPM31510 on Mitochondrial Energetics in Older Adults With Sarcopenia
Acronym: COQ10
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug manufacturing update. Study site will proceed with study in future.
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1665113
Record Dates: First submitted 2021-07-13; First posted 2021-08-10 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomized, parallel arm trial in which the supplementation with oral BPM 31510 or placebo will be blind.
Masking Description: Randomized, parallel arm trial in which the supplementation with oral BPM 31510 or placebo will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Older adults with sarcopenia (placebo) (Placebo Comparator)
  Interventions: Other: Placebo
- Older adults with sarcopenia (drug) (Active Comparator)
  Interventions: Drug: BPM31510

INTERVENTIONS:
Drug: BPM31510 — A total of 3200 mg of BPM 31510 or placebo will be self-administered daily by subjects before the morning, afternoon, and evening meals, with no fewer than 4 and no more than 6 hours elapsed between doses during the daytime.
  Arms: Older adults with sarcopenia (drug)
Other: Placebo — A total of 3200 mg of BPM 31510 or placebo will be self-administered daily by subjects before the morning, afternoon, and evening meals, with no fewer than 4 and no more than 6 hours elapsed between doses during the daytime.
  Arms: Older adults with sarcopenia (placebo)

SUMMARY:
This study is being done to gather data on whether oral supplementation of CoQ10 is enriched in the blood and muscles in older adults with sarcopenia. This study involves 28 consecutive days of oral CoQ10 supplementation to explore changes in muscle strength, aerobic capacity and physical function with CoQ10 supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be male or female, ages 65 through 90 years of age.
2. Participant must be sedentary, defined as ≤ 1 structured intentional continuous exercise session (approximately 30 mins) per week.
3. Participant must be sarcopenic, defined as having a skeletal muscle mass index (SMI) of <7.25 kg/m2 for males or <5.67 kg/m2 for females via DEXA scan.
4. Participant states willingness to follow the protocol as described and will complete any forms needed throughout the study.
5. Participant has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.

Exclusion Criteria:

1. Inability and/or unwillingness to comply with the protocol as written
2. Participant has had a significant cardiovascular event (e.g., myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure; or participant has evidence of cardiovascular disease assessed during the ECG at screening. In the event of a positive stress test, participants are referred to their primary care physician. If the electrocardiogram (ECG) is determined to be a false positive, participant may be allowed to participate in study after confirmatory records obtained.
3. The presence of any condition which contraindicate moderate exercise and would result in the inability to comply with the protocol as written or would compromise participant safety or data integrity, will be considered on a case-by-case basis by the Principal investigator and the study physician.
4. Participant is actively pursuing weight loss and/or lifestyle changes.
5. History of gastrointestinal or intracranial hemorrhage.
6. History of stroke or cerebrovascular accident.
7. Participant has diabetes.
8. Weight stable -no gain/loss by self-report of ≥ 10 lbs in 6 months prior to screening
9. BMI 40.0 kg/m2
10. Untreated or poorly controlled hypertension (SBP 150, DBP 95), or hypotension (SBP 100 DBP 60)
11. Participant has untreated hyperthyroidism (TSH (0.5mIU/L) or untreated hypothyroidism (TSH 10mIU/L).
12. Participant has current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months prior to screening visit.
13. Participant is currently taking anti-inflammatory medication or has had anti-inflammatory medication within 1 week prior to screening (including over the counter formulations, e.g., Aleve, Motrin, ibuprofen, naproxen, low dose aspirin).
14. Participant has had surgery requiring > 2 days of hospitalization in the last 1 month prior to screening visit.
15. Participant has an active malignancy or autoimmune disease.
16. Participant has current significantly impaired liver function in the opinion of the study Medical Investigator (mild asymptomatic fatty liver is acceptable), or hepatic enzyme tests are ≥ 2.5 times normal limit.
17. Participant has a chronic, contagious, or infectious diseases, such as active tuberculosis, Hepatitis B or C, or HIV, per self-report.
18. Participant currently has uncontrolled severe diarrhea, nausea or vomiting.
19. Participant has an obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome or other forms of gastrointestinal disease such as stage III or above gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis and bariatric surgery.
20. Participant has a mini-Mental State Examination score < 21.
21. Unable to participate in DXA assessments due to physical limitations of equipment tolerances (e.g., DXA 450-pound weight limit), claustrophobia, or based on Investigator's judgment at screening.
22. Participant has a sensitivity or allergy to lidocaine.
23. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.
24. Participant has peripheral vascular disease.
25. Participant has proteinuria defined as > 1+; approximately 30 mg/dl.
26. Clinically significant abnormality on ECG

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of skeletal muscle | Following 28 days of treatment
  We will evaluate changes in mitochondrial function (respiration) on permeabilized skeletal muscle fiber bundles obtained from biopsies of the vastus lateralis and blood draws, respectively. Blood and muscle biospecimens will also be obtained for multi-omics analysis.
Measurement of platelet CoQ10 level | Following 28 days of treatment
  We will evaluate changes in mitochondrial function (respiration) on cells (platelets) obtained from biopsies of the vastus lateralis and blood draws, respectively. Blood and muscle biospecimens will also be obtained for multi-omics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coen, PhD, Principal Investigator — AdventHealth Translational Research Institute
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States